CLINICAL TRIAL: NCT00913627
Title: Ibuprofen 600 Mg Extended Release (er) Single-dose Dental Pain Study
Brief Title: Study Evaluating Ibuprofen 600 mg Extended Release (ER) For Dental Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK-09-07; B4371001 (Other: Alias Study Number)
Record Dates: First submitted 2009-05-29; First posted 2009-06-04 (Estimated); Results first posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-02

CONDITIONS: Pain
Keywords: Extended-release; ibuprofen
MeSH Terms: conditions — Pain | interventions — Ibuprofen; Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): 1 x 600 mg ibuprofen IR/ER-roller compaction caplet
  Interventions: Drug: ibuprofen
- 2 (Experimental): 1 x 600 mg ibuprofen IR/ER-Wet granulation caplet
  Interventions: Drug: ibuprofen
- 3 (Active Comparator): 1x 220 mg naproxen sodium (Aleve caplet)
  Interventions: Drug: naproxen
- 4 (Placebo Comparator): 1 x placebo caplet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ibuprofen
  Arms: 1
Drug: ibuprofen
  Arms: 2
Drug: naproxen
  Arms: 3
Drug: Placebo
  Arms: 4

SUMMARY:
The purpose of this study is to assess the efficacy and safety of a single dose of an ibuprofen 600 mg extended release formulation in post-operative dental pain. There is concern that the manufacturing process may affect the performance characteristics of the selected prototype. Therefore, two formulations of this prototype manufactured by two different processes, [roller compaction] and [wet granulation] will be included in this study. The preferred prototype manufactured by two different methods will be compared to placebo and each other. This study will also characterize the pharmacokinetic/pharmacodynamic relationship with these formulations.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA:

* Males and females 16 to 40 years of age.
* Outpatients who undergo surgical extraction of 1-2 third molars, one of which must be a partial or full bony mandibular impaction and have moderate to severe post-operative pain (confirmed by a VAS score of at least 50 mm on a 100 mm VAS) following surgical extraction;
* Use of only the following preoperative medication(s)/anesthetic(s): short-acting local anesthetic (mepivacaine or lidocaine) with or without vasoconstrictor, nitrous oxide, and/or midazolam;
* Reliable, cooperative, and of adequate intelligence to record the requested information on the analgesic questionnaire form;
* Examined by the attending dentist or physician and medically cleared to participate in the study;
* In general good health and have no contraindications to the study medication.

Exclusion Criteria:

EXCLUSION CRITERIA:

* Pregnancy, as verified by a urine-based pregnancy test, or breast feeding;
* Presence of a serious medical condition (e.g., poorly controlled hypertension, poorly controlled diabetes, significantly impaired cardiac, renal or hepatic function, poorly-controlled hyper- or hypothyroidism);
* Use of a prescription or nonprescription drug with which the administration of ibuprofen or any other NSAID is contraindicated;
* Use of a bisphosphonate (e.g., risedronate [Actonel], alendronate [Fosamax], or ibandronate [Boniva]) in the past 5-years;
* Acute localized dentalveolar infection at the time of surgery that could confound the post-surgical evaluation;
* Females who are of child-bearing potential, or post-menopausal for less than 2 years and not using a medically approved method of contraception (i.e., oral, transdermal, or implanted contraceptives, intrauterine device, diaphragm, condom, abstinence, or surgical sterility), or females who test positive on a urine-based pregnancy test;
* Presence or history (within 2 years of enrollment) of bleeding disorder(s) or peptic ulcer disease;
* History of alcoholism (i.e., on average, consumes 3 or more alcoholic drinks per day) or substance abuse within the last year, or is currently abusing alcohol or other mood-altering drugs (e.g., cannabis). Patients who are taking CNS or other psychotropic drugs (including St. John's Wort, or any other nutritional supplement known to have psychotropic effects) may be enrolled if they have been on stable doses of medication for at least 2 months, will maintain this dose throughout the study, and their condition is judged by the Principal Investigator to be well-controlled;
* Habituation to analgesic drugs (i.e., routine use of oral analgesics 5 or more times per week)
* History of allergic reaction (e.g., asthma, rhinitis, swelling, shock, or hives) to ibuprofen, naproxen, aspirin, or to any other NSAID; or to codeine, hydrocodone, or acetaminophen, or to their combinations;
* Prior use of any type of analgesic or NSAID five half-lives of that drug or less before taking the first dose of study medication, except for pre-anesthetic medication and anesthesia for the procedure;
* Ingestion of any caffeine-containing beverages, chocolate, or alcohol 4 hours or less before taking the first dose of study medication;
* The subject has taken an investigational product or participated in an investigational trial within 30 days of study enrollment;
* The subject has previously participated in this study;
* The subject is a member of the study site staff directly involved with the study, an employee of the Sponsor, or a relative of study site personnel directly involved with the study.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 196 (Actual)
Dates: Start 2009-05-07 (Actual); Primary Completion 2009-08-01 (Actual); Study Completion 2009-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Jean Brown Research Center, Salt Lake City, Utah, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=AK-09-07&StudyName=Study%20Evaluating%20Ibuprofen%20600%20mg%20Extended%20Release%20%28ER%29%20For%20Dental%20Pain

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching placebo immediate release/extended release (IE/ER) caplet on day of surgery
- Ibuprofen IR/ER (Roller Compaction): Ibuprofen 600 milligram (mg) IR/ER-roller compaction (IR/ER-RC): one 600 mg active caplet on day of surgery
- Ibuprofen IR/ER (Wet Granulation): Ibuprofen 600 mg IR/ER-Wet Granulation (IR/ER-WG): one 600 mg active caplet on day of surgery
- Naproxen: Naproxen 220 mg (Aleve) caplet: one 220 mg active caplet on day of surgery
Period: Overall Study
Arm/Group | Placebo | Ibuprofen IR/ER (Roller Compaction) | Ibuprofen IR/ER (Wet Granulation) | Naproxen
Started | 29 | 53 | 56 | 58
Completed | 29 | 53 | 56 | 58
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ibuprofen IR/ER (Roller Compaction) | Ibuprofen IR/ER (Wet Granulation) | Naproxen | Total
Number analyzed (Participants) | 29 | 53 | 56 | 58 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.1 (2.1) | 18.6 (2.4) | 18.7 (2.7) | 18.3 (2.6) | 18.5 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 22 | 23 | 24 | 81
  Male | 17 | 31 | 33 | 34 | 115
Pain severity [Number; unit: participants] — A 4-point categorical pain intensity rating scale was used to rate the severity of baseline pain in response to the query, " My starting pain is:" Range of scale: None, Mild, Moderate, Severe. A baseline pain intensity score of at least moderate was required for study enrollment.
  participants
    Moderate | 18 | 29 | 33 | 34 | 114
    Severe | 11 | 24 | 23 | 24 | 82
Pain intensity [Mean (Standard Deviation); unit: mm] — Visual Analogue Scale (VAS) rated baseline pain intensity. Participants asked to "Draw a single vertical line on the scale that shows how much pain you have at this time." Scores measured to nearest millimeter (mm), ranged from 0 to 100 mm. Minimum 50 mm score required to verify participant had at least moderate pain at baseline.
  mm | 73.90 (11.60) | 77.06 (13.23) | 74.80 (12.40) | 75.12 (12.30) | 75.37 (12.44)

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Sum of Pain Intensity Difference Score From 0 to 12 Hours (SPID 0-12)
Description: Pain intensity difference (PID) score based on 4-point categorical pain intensity rating scale. Participants asked, "How much pain do you have at this time?" Range of scale: None (0), Mild (1), Moderate (2), Severe (3). SPID derived by adding the time-weighted sums of PID scores over the time interval. Scores could range from -12 to 36 where higher positive values indicated improvement (decrease in pain intensity).
Time Frame: Baseline (0 hour) to 12 hours post dose
Population: Intent-To-Treat (ITT) population: randomized participants who dosed with study product and provided a baseline pain severity assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen IR/ER (Roller Compaction) | Ibuprofen IR/ER (Wet Granulation) | Naproxen
Number analyzed (Participants) | 29 | 53 | 56 | 58
units on a scale | 0.05 (9.22) | 16.87 (9.35) | 17.34 (10.54) | 12.66 (10.02)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline pain severity rating (PSR) and gender; Mean Difference (Final Values) = 16.16, 95% CI 2-sided [12.13 to 20.19]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline pain severity rating (PSR) and gender; Mean Difference (Final Values) = 17.00, 95% CI 2-sided [13.02 to 20.99]
Statistical Analysis 3: Comparison: Placebo vs Naproxen; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline pain severity rating (PSR) and gender; Mean Difference (Final Values) = 12.30, 95% CI 2-sided [8.33 to 16.26]

2. Primary Outcome: Time-weighted Sum of Pain Intensity Difference Score From 8 to 12 Hours (SPID 8-12)
Description: PID score based on 4-point categorical pain intensity rating scale. Participants asked, "How much pain do you have at this time?" Range of scale: None (0), Mild (1), Moderate (2), Severe (3). SPID score derived by adding the time-weighted sums of PID scores over the time interval. Scores could range from -4 to 12 where higher positive values indicated improvement (decrease in pain intensity).
Time Frame: 8 to 12 hours post dose
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen IR/ER (Roller Compaction) | Ibuprofen IR/ER (Wet Granulation) | Naproxen
Number analyzed (Participants) | 29 | 53 | 56 | 58
units on a scale | -0.03 (4.05) | 6.57 (4.44) | 7.14 (5.24) | 5.14 (5.02)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 6.34, 95% CI 2-sided [4.30 to 8.38]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 7.06, 95% CI 2-sided [5.05 to 9.08]
Statistical Analysis 3: Comparison: Placebo vs Naproxen; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 5.05, 95% CI 2-sided [3.04 to 7.06]

3. Secondary Outcome: Time to First Perceptible Pain Relief
Description: Time to first perceptible relief (confirmed by meaningful relief) was defined as the elapsed time from dosing until the participant depresses the first stopwatch labelled "first perceptible relief", if the participant also depressed the second stopwatch labelled as "meaningful relief" by 6 hours. If the confirmation was not achieved, the participant was censored at 6 hours. Perceptible relief defined as when participant first begins to feel any pain relieving effect whatsoever of the drug. Does not necessarily mean the participant feels completely better, but when the participant first feels any difference in the pain he/she has currently.
Time Frame: Baseline to 6 hours
Population: ITT population
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Ibuprofen IR/ER (Roller Compaction) | Ibuprofen IR/ER (Wet Granulation) | Naproxen
Number analyzed (Participants) | 29 | 53 | 56 | 58
minutes | NA [NA to NA] — Data was not available as median time to onset of first perceptible pain relief was greater than (>) 360 minutes for placebo group. | 29.4 [23.3 to 35.3] | 29.4 [26.1 to 36.2] | 32.1 [29.5 to 58.0]

4. Secondary Outcome: Time to Treatment Failure
Description: Time to first rescue medication or discontinuation due to lack of efficacy
Time Frame: Baseline to 24 hours
Population: ITT population
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | Ibuprofen IR/ER (Roller Compaction) | Ibuprofen IR/ER (Wet Granulation) | Naproxen
Number analyzed (Participants) | 29 | 53 | 56 | 58
hours | 1.7 [1.7 to 2.2] | NA [NA to NA] — Data was not available as median time to treatment failure was greater than (>) 24 hours for Ibuprofen IR/ER (roller compaction)group. | NA [NA to NA] — Data was not available as median time to treatment failure was greater than (>) 24 hours for Ibuprofen IR/ER (wet granulation)group. | NA [NA to NA] — Data was not available as median time to treatment failure was greater than (>) 24 hours for Naproxen group.

5. Secondary Outcome: Percentage of Participants With Treatment Failure
Description: Treatment failure defined as use of rescue medication or discontinuation due to lack of efficacy.
Time Frame: 8, 9, 10, 11, and 12 hours
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ibuprofen IR/ER (Roller Compaction) | Ibuprofen IR/ER (Wet Granulation) | Naproxen
Number analyzed (Participants) | 29 | 53 | 56 | 58
percentage of participants
  8 hours | 82.8 | 11.3 | 12.5 | 24.1
  9 hours | 82.8 | 11.3 | 12.5 | 25.9
  10 hours | 82.8 | 17.0 | 12.5 | 27.6
  11 hours | 82.8 | 20.8 | 14.3 | 27.6
  12 hours | 82.8 | 20.8 | 17.9 | 32.8
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 8 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; Cochran-Mantel-Haenszel (CMH) = -72.19, 95% CI 2-sided [-88.56 to -55.83] — CMH adjusted proportions
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 8 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; Cochran-Mantel-Haenszel (CMH) = -70.72, 95% CI 2-sided [-87.14 to -54.30] — CMH adjusted proportions
Statistical Analysis 3: Comparison: Placebo vs Naproxen; 8 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; Cochran-Mantel-Haenszel (CMH) = -59.60, 95% CI 2-sided [-76.94 to -42.27] — CMH adjusted proportions
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 9 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; Cochran-Mantel-Haenszel (CMH) = -72.19, 95% CI 2-sided [-88.56 to -55.83] — CMH adjusted proportions
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 9 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; Cochran-Mantel-Haenszel (CMH) = -70.72, 95% CI 2-sided [-87.14 to -54.30] — CMH adjusted proportions
Statistical Analysis 6: Comparison: Placebo vs Naproxen; 9 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; Cochran-Mantel-Haenszel (CMH) = -57.79, 95% CI 2-sided [-75.43 to -40.16] — CMH adjusted proportions
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 10 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; Cochran-Mantel-Haenszel (CMH) = -66.79, 95% CI 2-sided [-83.98 to -49.60] — CMH adjusted proportions
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 10 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; Cochran-Mantel-Haenszel (CMH) = -70.72, 95% CI 2-sided [-87.14 to -54.30] — CMH adjusted proportions
Statistical Analysis 9: Comparison: Placebo vs Naproxen; 10 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; Cochran-Mantel-Haenszel (CMH) = -55.98, 95% CI 2-sided [-73.85 to -38.11] — CMH adjusted proportions
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 11 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = -63.44, 95% CI 2-sided [-80.82 to -46.06]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 11 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = -68.88, 95% CI 2-sided [-85.63 to -54.14]
Statistical Analysis 12: Comparison: Placebo vs Naproxen; 11 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = -55.98, 95% CI 2-sided [-73.85 to -38.11]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 12 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = -63.44, 95% CI 2-sided [-80.82 to -46.06]
Statistical Analysis 14: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 12 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = -65.28, 95% CI 2-sided [-82.49 to -48.07]
Statistical Analysis 15: Comparison: Placebo vs Naproxen; 12 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = -50.77, 95% CI 2-sided [-69.09 to -32.45]

6. Secondary Outcome: Time-weighted Sum of Pain Intensity Difference From 0 to 4 Hours (SPID 0-4) and 4 to 8 Hours (SPID 4-8)
Description: Time-weighted sum of PID score. PID based on 4-point categorical pain intensity rating scale. Participants asked, "How much pain do you have at this time?" Range of scale: None (0), Mild (1), Moderate (2), Severe (3). SPID score derived by adding the time-weighted sums of PID scores over the time interval. Scores could range from -4 to 12 where higher positive values indicated improvement (decrease in pain intensity).
Time Frame: 0 to 4 hours and 4 to 8 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen IR/ER (Roller Compaction) | Ibuprofen IR/ER (Wet Granulation) | Naproxen
Number analyzed (Participants) | 29 | 53 | 56 | 58
units on a scale
  SPID 0-4 | -0.12 (2.57) | 5.44 (3.21) | 5.22 (2.90) | 3.96 (2.87)
  SPID 4-8 | 0.31 (4.57) | 8.15 (4.48) | 8.13 (4.76) | 5.95 (4.74)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); SPID 0-4; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR, and gender; Mean Difference (Final Values) = 5.34, 95% CI 2-sided [4.18 to 6.51]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); SPID 0-4; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 5.25, 95% CI 2-sided [4.09 to 6.40]
Statistical Analysis 3: Comparison: Placebo vs Naproxen; SPID 0-4; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.98, 95% CI 2-sided [2.83 to 5.12]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); SPID 4-8; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 7.53, 95% CI 2-sided [5.63 to 9.43]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); SPID 4-8; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 7.68, 95% CI 2-sided [5.80 to 9.56]
Statistical Analysis 6: Comparison: Placebo vs Naproxen; SPID 4-8; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 5.49, 95% CI 2-sided [3.62 to 7.36]

7. Secondary Outcome: Time-weighted Sum of Pain Relief and Pain Intensity Difference Scores (SPRID)
Description: Time-weighted sum of PRID score where PRID=PID+PR. PID: 4-point categorical pain intensity difference scale, 0 (none) to 3 (severe), score derived by subtracting postdose score from baseline, ranged from -1 to 3. Baseline pain intensity score of at least 2 required for enrollment. Higher positive PID values = improvement. PR: 5-point categorical pain relief scale None (0), A Little (1), Some (2), A Lot (3) or Complete (4). SPRID 0-4, SPRID 4-8, and SRID 8-12 scores ranged from -4 to 28, SPRID 0-12 ranged from -12 to 84, higher scores = greater improvement.
Time Frame: 0 to 4 hours, 4 to 8 hours, 8 to 12 hours, and 0 to 12 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen IR/ER (Roller Compaction) | Ibuprofen IR/ER (Wet Granulation) | Naproxen
Number analyzed (Participants) | 29 | 53 | 56 | 58
units on a scale
  SPRID 0-4 | 1.78 (5.45) | 15.48 (6.60) | 15.12 (6.10) | 11.97 (6.51)
  SPRID 4-8 | 3.69 (10.63) | 23.21 (8.85) | 23.14 (10.12) | 17.71 (10.69)
  SPRID 8-12 | 3.00 (9.38) | 19.36 (9.94) | 20.73 (11.43) | 15.86 (11.56)
  SPRID 0-12 | 7.09 (21.00) | 48.76 (18.99) | 50.01 (22.32) | 38.45 (22.61)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); SPRID 0-4; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 13.47, 95% CI 2-sided [10.68 to 16.27]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); SPRID 0-4; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 13.24, 95% CI 2-sided [10.48 to 16.01]
Statistical Analysis 3: Comparison: Placebo vs Naproxen; SPRID 0-4; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 10.08, 95% CI 2-sided [7.33 to 12.83]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); SPRID 4-8; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 19.21, 95% CI 2-sided [14.71 to 23.71]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); SPRID 4-8; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 19.32, 95% CI 2-sided [14.86 to 23.78]
Statistical Analysis 6: Comparison: Placebo vs Naproxen; SPRID 4-8; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 13.87, 95% CI 2-sided [9.44 to 18.30]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); SPRID 8-12; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 16.18, 95% CI 2-sided [11.29 to 21.07]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); SPRID 8-12; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 17.65, 95% CI 2-sided [12.81 to 22.49]
Statistical Analysis 9: Comparison: Placebo vs Naproxen; SPRID 8-12; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 12.78, 95% CI 2-sided [7.97 to 17.59]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); SPRID 0-12; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 41.08, 95% CI 2-sided [31.48 to 50.69]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); SPRID 0-12; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 42.66, 95% CI 2-sided [33.15 to 52.17]
Statistical Analysis 12: Comparison: Placebo vs Naproxen; SPRID 0-12; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 31.08, 95% CI 2-sided [21.63 to 40.53]

8. Secondary Outcome: Time-weighted Sum of Pain Relief Scores (TOTPAR)
Description: TOTPAR based on 5-point categorical pain relief scale. Participants asked, "How much relief do you have from your starting pain?" Range of scale: None (0), A Little (1), Some (2), A Lot (3) or Complete (4). Higher scores indicated improvement (better pain relief). For time-weighted sum of pain relief scores from 0 to 4 hours (TOTPAR 0-4), from 4 to 8 hours (TOTPAR 4-8), and from 8 to 12 hours (TOTPAR 8-12): range of scores 0 (worst) to 16 (best). TOTPAR 0-12 range of scores 0 (worst) to 48 (best).
Time Frame: 0 to 4 hours, 4 to 8 hours, 8 to 12 hours, and 0 to 12 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen IR/ER (Roller Compaction) | Ibuprofen IR/ER (Wet Granulation) | Naproxen
Number analyzed (Participants) | 29 | 53 | 56 | 58
units on a scale
  TOTPAR 0-4 | 1.91 (3.25) | 10.04 (3.66) | 9.90 (3.51) | 8.01 (3.96)
  TOTPAR 4-8 | 3.38 (6.43) | 15.06 (4.76) | 15.02 (5.79) | 11.76 (6.35)
  TOTPAR 8-12 | 3.03 (5.75) | 12.79 (5.97) | 13.59 (6.61) | 10.72 (6.89)
  TOTPAR 0-12 | 7.04 (12.74) | 31.89 (10.67) | 32.67 (12.74) | 25.79 (13.48)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); TOTPAR 0-4; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 8.13, 95% CI 2-sided [6.45 to 9.80]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); TOTPAR 0-4; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 7.99, 95% CI 2-sided [6.34 to 9.65]
Statistical Analysis 3: Comparison: Placebo vs Naproxen; TOTPAR 0-4; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 6.11, 95% CI 2-sided [4.46 to 7.75]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); TOTPAR 4-8; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 11.68, 95% CI 2-sided [9.02 to 14.34]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); TOTPAR 4-8; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 11.64, 95% CI 2-sided [9.01 to 14.27]
Statistical Analysis 6: Comparison: Placebo vs Naproxen; TOTPAR 4-8; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 8.38, 95% CI 2-sided [5.76 to 11.00]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); TOTPAR 8-12; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 9.84, 95% CI 2-sided [6.93 to 12.75]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); TOTPAR 8-12; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 10.59, 95% CI 2-sided [7.71 to 13.46]
Statistical Analysis 9: Comparison: Placebo vs Naproxen; TOTPAR 8-12; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 7.73, 95% CI 2-sided [4.87 to 10.59]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); TOTPAR 0-12; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 24.93, 95% CI 2-sided [19.24 to 30.61]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); TOTPAR 0-12; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 25.66, 95% CI 2-sided [20.03 to 31.28]
Statistical Analysis 12: Comparison: Placebo vs Naproxen; TOTPAR 0-12; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 18.78, 95% CI 2-sided [13.19 to 24.38]

9. Secondary Outcome: Percentage of Participants Achieving First Perceptible Relief Confirmed by Meaningful Relief
Description: The elapsed time from dosing until the participant indicated first perceptible relief, provided the participant also indicated achieving meaningful relief. Perceptible relief defined as when participant first begins to feel any pain-relieving effect whatsoever of the drug. Does not necessarily mean the participant feels completely better, but when the participant first feels any difference in the pain he/she currently has now.
Time Frame: 15, 30, 45, 60, 90, and 120 minutes and every 60 minutes up to 360 minutes
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ibuprofen IR/ER (Roller Compaction) | Ibuprofen IR/ER (Wet Granulation) | Naproxen
Number analyzed (Participants) | 29 | 53 | 56 | 58
percentage of participants
  15 minutes | 3.4 | 17.0 | 19.6 | 8.6
  30 minutes | 3.4 | 52.8 | 55.4 | 39.7
  45 minutes | 6.9 | 64.2 | 73.2 | 56.9
  60 minutes | 13.8 | 81.1 | 83.9 | 65.5
  90 minutes | 13.8 | 83.0 | 87.5 | 72.4
  120 minutes | 13.8 | 83.0 | 91.1 | 72.4
  180 minutes | 13.8 | 83.0 | 91.1 | 72.4
  240 minutes | 13.8 | 83.0 | 91.1 | 72.4
  300 minutes | 13.8 | 83.0 | 91.1 | 72.4
  360 minutes | 13.8 | 83.0 | 91.1 | 72.4
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 15 minutes; Test type: Superiority or Other; p = 0.080, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 13.31, 95% CI 2-sided [1.26 to 25.36]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 15 minutes; Test type: Superiority or Other; p = 0.043, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 16.39, 95% CI 2-sided [3.73 to 29.04]
Statistical Analysis 3: Comparison: Placebo vs Naproxen; 15 minutes; Test type: Superiority or Other; p = 0.354, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 5.39, 95% CI 2-sided [-4.62 to 15.40]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 30 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 48.65, 95% CI 2-sided [33.34 to 63.96]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 30 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 51.94, 95% CI 2-sided [37.15 to 66.73]
Statistical Analysis 6: Comparison: Placebo vs Naproxen; 30 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 36.80, 95% CI 2-sided [22.62 to 50.98]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 45 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 57.39, 95% CI 2-sided [41.20 to 73.57]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 45 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 66.67, 95% CI 2-sided [51.56 to 81.78]
Statistical Analysis 9: Comparison: Placebo vs Naproxen; 45 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 50.20, 95% CI 2-sided [34.20 to 66.21]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 60 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 67.64, 95% CI 2-sided [51.36 to 83.93]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 60 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 70.61, 95% CI 2-sided [55.16 to 86.05]
Statistical Analysis 12: Comparison: Placebo vs Naproxen; 60 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 51.85, 95% CI 2-sided [34.32 to 69.38]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 90 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 69.33, 95% CI 2-sided [53.33 to 85.33]
Statistical Analysis 14: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 90 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 74.21, 95% CI 2-sided [59.29 to 89.14]
Statistical Analysis 15: Comparison: Placebo vs Naproxen; 90 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 58.86, 95% CI 2-sided [41.88 to 75.84]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 120 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 69.33, 95% CI 2-sided [53.33 to 85.33]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 120 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 77.82, 95% CI 2-sided [63.57 to 92.06]
Statistical Analysis 18: Comparison: Placebo vs Naproxen; 120 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 58.86, 95% CI 2-sided [41.88 to 75.84]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 180 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 69.33, 95% CI 2-sided [53.33 to 85.33]
Statistical Analysis 20: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 180 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 77.82, 95% CI 2-sided [63.57 to 92.06]
Statistical Analysis 21: Comparison: Placebo vs Naproxen; 180 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 58.86, 95% CI 2-sided [41.88 to 75.84]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 240 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 69.33, 95% CI 2-sided [53.33 to 85.33]
Statistical Analysis 23: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 240 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 77.82, 95% CI 2-sided [63.57 to 92.06]
Statistical Analysis 24: Comparison: Placebo vs Naproxen; 240 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 58.86, 95% CI 2-sided [41.88 to 75.84]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 300 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 69.33, 95% CI 2-sided [53.33 to 85.33]
Statistical Analysis 26: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 300 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 77.82, 95% CI 2-sided [63.57 to 92.06]
Statistical Analysis 27: Comparison: Placebo vs Naproxen; 300 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 58.86, 95% CI 2-sided [41.88 to 75.84]
Statistical Analysis 28: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 360 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 69.33, 95% CI 2-sided [53.33 to 85.33]
Statistical Analysis 29: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 360 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 77.82, 95% CI 2-sided [63.57 to 92.06]
Statistical Analysis 30: Comparison: Placebo vs Naproxen; 360 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 58.86, 95% CI 2-sided [41.88 to 75.84]

10. Secondary Outcome: Time to Meaningful Pain Relief
Description: Participants evaluated the time to meaningful relief by depressing a second stopwatch at the moment they first began to experience meaningful relief, defined as relief from the pain that is considered meaningful to the participant.
Time Frame: Baseline to 6 hours
Population: ITT population
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Ibuprofen IR/ER (Roller Compaction) | Ibuprofen IR/ER (Wet Granulation) | Naproxen
Number analyzed (Participants) | 29 | 53 | 56 | 58
minutes | NA [NA to NA] — Median time to meaningful pain relief not achieved by more than 50 percent (%) of participants. | 59.7 [52.3 to 88.3] | 76.7 [56.5 to 99.3] | 84.1 [63.8 to 174.2]
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); Test type: Superiority or Other; p < 0.001, Proportional hazards regression — p-value adjusted for gender and categorical baseline pain severity; Hazard Ratio, log = 13.56, 95% CI 2-sided [4.85 to 37.89]

11. Secondary Outcome: Percentage of Participants Achieving Meaningful Pain Relief
Description: Participants evaluated the time to first perceptible pain relief by depressing a stopwatch at the moment they first began to experience perceptible relief and the time to meaningful relief by depressing a second stopwatch at the moment they first began to experience meaningful relief defined as relief from the pain that is considered meaningful to the participant.
Time Frame: 15, 30, 45, 60, 90, and 120 minutes and every 60 minutes up to 360 minutes
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ibuprofen IR/ER (Roller Compaction) | Ibuprofen IR/ER (Wet Granulation) | Naproxen
Number analyzed (Participants) | 29 | 53 | 56 | 58
percentage of participants
  15 minutes | 0.0 | 1.9 | 0.0 | 1.7
  30 minutes | 0.0 | 9.4 | 10.7 | 3.4
  45 minutes | 3.4 | 28.3 | 28.6 | 13.8
  60 minutes | 3.4 | 50.9 | 39.3 | 31.0
  90 minutes | 3.4 | 64.2 | 57.1 | 50.0
  120 minutes | 6.9 | 71.7 | 71.4 | 56.9
  180 minutes | 10.3 | 79.2 | 82.1 | 63.8
  240 minutes | 10.3 | 83.0 | 89.3 | 67.2
  300 minutes | 10.3 | 83.0 | 91.1 | 69.0
  360 minutes | 13.8 | 83.0 | 91.1 | 72.4
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 15 minutes; Test type: Superiority or Other; p = 0.434, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 2.03, 95% CI 2-sided [-1.95 to 6.02]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 15 minutes; Test type: Superiority or Other; Cochran-Mantel-Haenszel; CMH adjusted proportions = 0.00, 95% CI 2-sided [0.00 to 0.00]
Statistical Analysis 3: Comparison: Placebo vs Naproxen; 15 minutes; Test type: Superiority or Other; p = 0.469, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 1.78, 95% CI 2-sided [-1.71 to 5.27]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 30 minutes; Test type: Superiority or Other; p = 0.101, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 9.13, 95% CI 2-sided [1.33 to 16.93]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 30 minutes; Test type: Superiority or Other; p = 0.069, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 10.73, 95% CI 2-sided [2.54 to 18.91]
Statistical Analysis 6: Comparison: Placebo vs Naproxen; 30 minutes; Test type: Superiority or Other; p = 0.303, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 3.59, 95% CI 2-sided [-1.39 to 8.57]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 45 minutes; Test type: Superiority or Other; p = 0.008, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 24.58, 95% CI 2-sided [10.68 to 38.47]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 45 minutes; Test type: Superiority or Other; p = 0.007, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 25.31, 95% CI 2-sided [11.35 to 39.28]
Statistical Analysis 9: Comparison: Placebo vs Naproxen; 45 minutes; Test type: Superiority or Other; p = 0.129, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 10.62, 95% CI 2-sided [-0.68 to 21.92]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 60 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 47.72, 95% CI 2-sided [32.25 to 63.19]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 60 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 36.01, 95% CI 2-sided [21.24 to 50.78]
Statistical Analysis 12: Comparison: Placebo vs Naproxen; 60 minutes; Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 27.87, 95% CI 2-sided [13.93 to 41.81]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 90 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 61.01, 95% CI 2-sided [46.12 to 75.89]
Statistical Analysis 14: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 90 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 53.83, 95% CI 2-sided [38.85 to 68.80]
Statistical Analysis 15: Comparison: Placebo vs Naproxen; 90 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 46.74, 95% CI 2-sided [31.89 to 61.58]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 120 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 64.78, 95% CI 2-sided [49.37 to 80.18]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 120 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 64.80, 95% CI 2-sided [50.01 to 79.59]
Statistical Analysis 18: Comparison: Placebo vs Naproxen; 120 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 50.19, 95% CI 2-sided [34.27 to 66.11]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 180 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 68.59, 95% CI 2-sided [52.81 to 84.38]
Statistical Analysis 20: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 180 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 72.16, 95% CI 2-sided [57.05 to 87.26]
Statistical Analysis 21: Comparison: Placebo vs Naproxen; 180 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 53.47, 95% CI 2-sided [36.57 to 70.37]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 240 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 72.66, 95% CI 2-sided [57.48 to 87.84]
Statistical Analysis 23: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 240 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 79.36, 95% CI 2-sided [65.68 to 93.05]
Statistical Analysis 24: Comparison: Placebo vs Naproxen; 240 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 57.03, 95% CI 2-sided [40.46 to 73.60]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 300 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 72.66, 95% CI 2-sided [57.48 to 87.84]
Statistical Analysis 26: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 300 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 81.20, 95% CI 2-sided [67.91 to 94.49]
Statistical Analysis 27: Comparison: Placebo vs Naproxen; 300 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 58.84, 95% CI 2-sided [42.34 to 75.35]
Statistical Analysis 28: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 360 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 69.33, 95% CI 2-sided [53.33 to 85.33]
Statistical Analysis 29: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 360 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 77.82, 95% CI 2-sided [63.57 to 92.06]
Statistical Analysis 30: Comparison: Placebo vs Naproxen; 360 minutes; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value adjusted for baseline PSR and gender; CMH adjusted proportions = 58.86, 95% CI 2-sided [41.88 to 75.84]

12. Secondary Outcome: Participant Global Evaluation of Study Medication at 12 Hours
Description: Participant rated global evaluation of study medication; results reported by evaluation categories and included very poor (0), poor (1), fair (2), good (3), very good (4), and excellent (5).
Time Frame: 12 hours
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Placebo | Ibuprofen IR/ER (Roller Compaction) | Ibuprofen IR/ER (Wet Granulation) | Naproxen
Number analyzed (Participants) | 29 | 53 | 56 | 58
participants
  Very poor | 20 | 2 | 2 | 7
  Poor | 4 | 1 | 0 | 1
  Fair | 1 | 3 | 4 | 8
  Good | 2 | 11 | 9 | 18
  Very good | 2 | 20 | 28 | 15
  Excellent | 0 | 16 | 13 | 9
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value from CMH test with modified ridit scores, adjusted for baseline PSR and gender; Goodman-Kruskal Gamma Statistic = 0.93, 95% CI 2-sided [0.85 to 1.01]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value from CMH test with modified ridit scores, adjusted for baseline PSR and gender; Goodman-Kruskal Gamma Statistic = 0.95, 95% CI 2-sided [0.88 to 1.02]
Statistical Analysis 3: Comparison: Placebo vs Naproxen; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value from CMH test with modified ridit scores, adjusted for baseline PSR and gender; Goodman-Kruskal Gamma Statistic = 0.84, 95% CI 2-sided [0.70 to 0.98]

13. Secondary Outcome: Participant Global Evaluation of Study Medication at 24 Hours
Description: as for outcome 12
Time Frame: 24 hours
Population: ITT population; Number of participants analyzed (N)= participants with evaluable data
Measure: Number; unit: participants
Arm/Group | Placebo | Ibuprofen IR/ER (Roller Compaction) | Ibuprofen IR/ER (Wet Granulation) | Naproxen
Number analyzed (Participants) | 29 | 52 | 56 | 58
participants
  Very poor | 20 | 2 | 2 | 7
  Poor | 4 | 1 | 0 | 1
  Fair | 1 | 2 | 3 | 4
  Good | 3 | 14 | 10 | 17
  Very good | 1 | 17 | 23 | 19
  Excellent | 0 | 16 | 18 | 10
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value from CMH test with modified ridit scores, adjusted for baseline PSR and gender; Goodman-Kruskal Gamma Statistic = 0.93, 95% CI 2-sided [0.85 to 1.01]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value from CMH test with modified ridit scores, adjusted for baseline PSR and gender; Goodman-Kruskal Gamma Statistic = 0.96, 95% CI 2-sided [0.91 to 1.01]
Statistical Analysis 3: Comparison: Placebo vs Naproxen; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value from CMH test with modified ridit scores, adjusted for baseline PSR and gender; Goodman-Kruskal Gamma Statistic = 0.89, 95% CI 2-sided [0.79 to 0.99]

14. Secondary Outcome: Pain Intensity Difference (PID) Score
Description: PID based on 4-point categorical pain intensity rating scale. Participants asked, "How much pain do you have at this time?" Range of scale: None (0), Mild (1), Moderate (2), Severe (3). PID score derived by subtracting postdose score from baseline score and could range from -1 to 3. A baseline pain intensity score of at least 2 was required for study enrollment. Higher positive PID values indicated greater improvement (decrease in pain intensity).
Time Frame: 15, 30, 45, 60, 90 minutes and 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 16, and 24 hours
Population: ITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen IR/ER (Roller Compaction) | Ibuprofen IR/ER (Wet Granulation) | Naproxen
Number analyzed (Participants) | 29 | 53 | 56 | 58
units on a scale
  15 minutes | -0.14 (0.44) | 0.09 (0.45) | 0.09 (0.35) | 0.05 (0.22)
  30 minutes | -0.14 (0.52) | 0.40 (0.69) | 0.34 (0.64) | 0.29 (0.53)
  45 minutes | -0.10 (0.56) | 0.77 (0.89) | 0.70 (0.78) | 0.53 (0.60)
  60 minutes | -0.10 (0.62) | 0.94 (0.99) | 1.00 (0.81) | 0.81 (0.76)
  90 minutes | -0.07 (0.59) | 1.25 (1.02) | 1.29 (0.87) | 1.05 (0.80)
  2 hours: number analyzed (Participants) | 13 | 51 | 54 | 53
  2 hours | 0.00 (0.65) | 1.51 (0.97) | 1.48 (0.91) | 1.05 (0.83)
  3 hours: number analyzed (Participants) | 8 | 51 | 53 | 52
  3 hours | 0.00 (0.85) | 1.70 (0.97) | 1.64 (0.88) | 1.24 (0.94)
  4 hours: number analyzed (Participants) | 7 | 51 | 51 | 51
  4 hours | 0.03 (0.94) | 1.81 (0.92) | 1.66 (0.94) | 1.24 (0.98)
  5 hours: number analyzed (Participants) | 7 | 51 | 51 | 50
  5 hours | 0.07 (0.92) | 1.74 (0.94) | 1.68 (0.97) | 1.22 (1.04)
  6 hours: number analyzed (Participants) | 7 | 51 | 51 | 47
  6 hours | 0.07 (0.92) | 1.62 (0.99) | 1.66 (0.98) | 1.22 (1.04)
  7 hours: number analyzed (Participants) | 7 | 51 | 51 | 47
  7 hours | 0.07 (0.92) | 1.51 (0.97) | 1.64 (0.98) | 1.12 (1.01)
  8 hours: number analyzed (Participants) | 7 | 49 | 50 | 46
  8 hours | 0.07 (0.92) | 1.47 (0.91) | 1.48 (1.06) | 1.14 (1.00)
  9 hours: number analyzed (Participants) | 7 | 49 | 50 | 45
  9 hours | 0.00 (0.80) | 1.34 (0.94) | 1.41 (1.06) | 1.00 (1.03)
  10 hours: number analyzed (Participants) | 7 | 47 | 50 | 44
  10 hours | -0.03 (0.78) | 1.26 (0.96) | 1.45 (1.11) | 1.02 (1.05)
  11 hours: number analyzed (Participants) | 7 | 46 | 49 | 44
  11 hours | -0.03 (0.82) | 1.23 (0.97) | 1.43 (1.11) | 1.03 (1.11)
  12 hours: number analyzed (Participants) | 7 | 46 | 47 | 41
  12 hours | -0.03 (0.82) | 1.26 (0.96) | 1.38 (1.09) | 0.95 (1.08)
  13 hours: number analyzed (Participants) | 6 | 43 | 44 | 41
  13 hours | 0.00 (0.85) | 1.25 (1.02) | 1.23 (1.14) | 0.95 (1.03)
  14 hours: number analyzed (Participants) | 6 | 41 | 43 | 40
  14 hours | 0.03 (0.91) | 1.15 (1.10) | 1.18 (1.15) | 0.93 (1.06)
  16 hours: number analyzed (Participants) | 6 | 39 | 39 | 38
  16 hours | -0.03 (0.82) | 1.08 (1.05) | 1.02 (1.10) | 0.95 (1.07)
  24 hours: number analyzed (Participants) | 2 | 4 | 1 | 2
  24 hours | 0.07 (1.00) | 0.89 (1.01) | 0.91 (1.13) | 0.97 (1.08)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 15 minutes; Test type: Superiority or Other; p = 0.008, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [0.06 to 0.38]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 15 minutes; Test type: Superiority or Other; p = 0.007, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [0.06 to 0.38]
Statistical Analysis 3: Comparison: Placebo vs Naproxen; 15 minutes; Test type: Superiority or Other; p = 0.024, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [0.02 to 0.34]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 30 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [0.24 to 0.78]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 30 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [0.20 to 0.73]
Statistical Analysis 6: Comparison: Placebo vs Naproxen; 30 minutes; Test type: Superiority or Other; p = 0.002, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [0.16 to 0.68]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 45 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.85, 95% CI 2-sided [0.52 to 1.17]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 45 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.79, 95% CI 2-sided [0.47 to 1.11]
Statistical Analysis 9: Comparison: Placebo vs Naproxen; 45 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.62, 95% CI 2-sided [0.30 to 0.94]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 60 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.01, 95% CI 2-sided [0.65 to 1.37]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 60 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.09, 95% CI 2-sided [0.73 to 1.44]
Statistical Analysis 12: Comparison: Placebo vs Naproxen; 60 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.90, 95% CI 2-sided [0.54 to 1.25]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 90 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.26, 95% CI 2-sided [0.90 to 1.63]
Statistical Analysis 14: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 90 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.33, 95% CI 2-sided [0.97 to 1.69]
Statistical Analysis 15: Comparison: Placebo vs Naproxen; 90 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.10, 95% CI 2-sided [0.74 to 1.45]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 2 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.45, 95% CI 2-sided [1.09 to 1.82]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 2 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.46, 95% CI 2-sided [1.10 to 1.82]
Statistical Analysis 18: Comparison: Placebo vs Naproxen; 2 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.03, 95% CI 2-sided [0.67 to 1.38]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 3 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.63, 95% CI 2-sided [1.26 to 2.00]
Statistical Analysis 20: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 3 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.61, 95% CI 2-sided [1.25 to 1.98]
Statistical Analysis 21: Comparison: Placebo vs Naproxen; 3 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.21, 95% CI 2-sided [0.85 to 1.57]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 4 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.71, 95% CI 2-sided [1.33 to 2.08]
Statistical Analysis 23: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 4 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.60, 95% CI 2-sided [1.23 to 1.97]
Statistical Analysis 24: Comparison: Placebo vs Naproxen; 4 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.17, 95% CI 2-sided [0.81 to 1.54]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 5 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.60, 95% CI 2-sided [1.20 to 2.00]
Statistical Analysis 26: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 5 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.58, 95% CI 2-sided [1.19 to 1.98]
Statistical Analysis 27: Comparison: Placebo vs Naproxen; 5 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.12, 95% CI 2-sided [0.73 to 1.52]
Statistical Analysis 28: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 6 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.49, 95% CI 2-sided [1.08 to 1.90]
Statistical Analysis 29: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 6 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.56, 95% CI 2-sided [1.16 to 1.97]
Statistical Analysis 30: Comparison: Placebo vs Naproxen; 6 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.13, 95% CI 2-sided [0.72 to 1.53]
Statistical Analysis 31: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 7 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.38, 95% CI 2-sided [0.97 to 1.79]
Statistical Analysis 32: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 7 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.55, 95% CI 2-sided [1.14 to 1.95]
Statistical Analysis 33: Comparison: Placebo vs Naproxen; 7 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.02, 95% CI 2-sided [0.62 to 1.43]
Statistical Analysis 34: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 8 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.35, 95% CI 2-sided [0.93 to 1.77]
Statistical Analysis 35: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 8 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.39, 95% CI 2-sided [0.97 to 1.81]
Statistical Analysis 36: Comparison: Placebo vs Naproxen; 8 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.04, 95% CI 2-sided [0.63 to 1.46]
Statistical Analysis 37: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 9 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.29, 95% CI 2-sided [0.87 to 1.71]
Statistical Analysis 38: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 9 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.39, 95% CI 2-sided [0.97 to 1.81]
Statistical Analysis 39: Comparison: Placebo vs Naproxen; 9 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.98, 95% CI 2-sided [0.56 to 1.39]
Statistical Analysis 40: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 10 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.25, 95% CI 2-sided [0.82 to 1.68]
Statistical Analysis 41: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 10 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.46, 95% CI 2-sided [1.03 to 1.89]
Statistical Analysis 42: Comparison: Placebo vs Naproxen; 10 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.03, 95% CI 2-sided [0.60 to 1.45]
Statistical Analysis 43: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 11 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.21, 95% CI 2-sided [0.77 to 1.64]
Statistical Analysis 44: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 11 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.44, 95% CI 2-sided [1.00 to 1.87]
Statistical Analysis 45: Comparison: Placebo vs Naproxen; 11 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.04, 95% CI 2-sided [0.61 to 1.48]
Statistical Analysis 46: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 12 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.25, 95% CI 2-sided [0.81 to 1.68]
Statistical Analysis 47: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 12 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.39, 95% CI 2-sided [0.96 to 1.82]
Statistical Analysis 48: Comparison: Placebo vs Naproxen; 12 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.96, 95% CI 2-sided [0.53 to 1.39]
Statistical Analysis 49: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 13 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.20, 95% CI 2-sided [0.75 to 1.64]
Statistical Analysis 50: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 13 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.21, 95% CI 2-sided [0.77 to 1.65]
Statistical Analysis 51: Comparison: Placebo vs Naproxen; 13 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.93, 95% CI 2-sided [0.49 to 1.36]
Statistical Analysis 52: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 14 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.07, 95% CI 2-sided [0.60 to 1.53]
Statistical Analysis 53: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 14 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.12, 95% CI 2-sided [0.66 to 1.58]
Statistical Analysis 54: Comparison: Placebo vs Naproxen; 14 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.87, 95% CI 2-sided [0.42 to 1.33]
Statistical Analysis 55: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 16 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.06, 95% CI 2-sided [0.61 to 1.51]
Statistical Analysis 56: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 16 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.03, 95% CI 2-sided [0.58 to 1.48]
Statistical Analysis 57: Comparison: Placebo vs Naproxen; 16 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.96, 95% CI 2-sided [0.52 to 1.40]
Statistical Analysis 58: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 24 hours; Test type: Superiority or Other; p = 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.77, 95% CI 2-sided [0.31 to 1.24]
Statistical Analysis 59: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 24 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.82, 95% CI 2-sided [0.36 to 1.28]
Statistical Analysis 60: Comparison: Placebo vs Naproxen; 24 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.88, 95% CI 2-sided [0.42 to 1.33]

15. Secondary Outcome: Pain Relief (PR) Score
Description: PR score based on 5-point categorical pain relief scale. Participants asked, "How much relief do you have from your starting pain?" Range of scale: None [0], A Little [1], Some [2], A Lot [3] or Complete [4]. Higher scores indicated improvement (better pain relief).
Time Frame: 15, 30, 45, 60, 90 minutes and 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 16, and 24 hours
Population: ITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen IR/ER (Roller Compaction) | Ibuprofen IR/ER (Wet Granulation) | Naproxen
Number analyzed (Participants) | 29 | 53 | 56 | 58
units on a scale
  15 minutes | 0.07 (0.26) | 0.36 (0.71) | 0.29 (0.56) | 0.28 (0.64)
  30 minutes | 0.21 (0.62) | 1.02 (0.99) | 0.82 (0.86) | 0.79 (0.91)
  45 minutes | 0.31 (0.66) | 1.72 (1.21) | 1.55 (1.17) | 1.21 (1.07)
  60 minutes | 0.41 (0.68) | 2.04 (1.27) | 1.98 (1.17) | 1.67 (1.19)
  90 minutes | 0.41 (0.73) | 2.40 (1.29) | 2.50 (1.16) | 2.09 (1.19)
  2 hours: number analyzed (Participants) | 13 | 51 | 54 | 53
  2 hours | 0.55 (0.91) | 2.66 (1.21) | 2.77 (1.14) | 2.24 (1.19)
  3 hours: number analyzed (Participants) | 8 | 51 | 53 | 52
  3 hours | 0.55 (1.15) | 3.06 (1.05) | 3.04 (1.09) | 2.43 (1.20)
  4 hours: number analyzed (Participants) | 7 | 51 | 51 | 51
  4 hours | 0.62 (1.27) | 3.17 (0.98) | 3.07 (1.13) | 2.43 (1.27)
  5 hours: number analyzed (Participants) | 7 | 51 | 51 | 50
  5 hours | 0.66 (1.29) | 3.13 (0.98) | 3.07 (1.19) | 2.36 (1.37)
  6 hours: number analyzed (Participants) | 7 | 51 | 51 | 47
  6 hours | 0.72 (1.36) | 2.98 (1.07) | 3.09 (1.16) | 2.40 (1.40)
  7 hours: number analyzed (Participants) | 7 | 51 | 51 | 47
  7 hours | 0.72 (1.36) | 2.94 (1.01) | 3.02 (1.20) | 2.29 (1.39)
  8 hours: number analyzed (Participants) | 7 | 49 | 50 | 46
  8 hours | 0.66 (1.26) | 2.83 (1.12) | 2.77 (1.33) | 2.28 (1.42)
  9 hours: number analyzed (Participants) | 7 | 49 | 50 | 45
  9 hours | 0.66 (1.23) | 2.55 (1.31) | 2.77 (1.32) | 2.16 (1.41)
  10 hours: number analyzed (Participants) | 7 | 47 | 50 | 44
  10 hours | 0.59 (1.15) | 2.51 (1.32) | 2.77 (1.36) | 2.14 (1.41)
  11 hours: number analyzed (Participants) | 7 | 46 | 49 | 44
  11 hours | 0.59 (1.21) | 2.47 (1.32) | 2.71 (1.37) | 2.17 (1.46)
  12 hours: number analyzed (Participants) | 7 | 46 | 47 | 41
  12 hours | 0.55 (1.18) | 2.43 (1.38) | 2.57 (1.45) | 1.98 (1.52)
  13 hours: number analyzed (Participants) | 6 | 43 | 44 | 41
  13 hours | 0.62 (1.27) | 2.43 (1.46) | 2.39 (1.53) | 2.03 (1.50)
  14 hours: number analyzed (Participants) | 6 | 41 | 43 | 40
  14 hours | 0.66 (1.34) | 2.28 (1.49) | 2.27 (1.60) | 2.03 (1.57)
  16 hours: number analyzed (Participants) | 6 | 39 | 39 | 38
  16 hours | 0.59 (1.27) | 2.15 (1.47) | 2.00 (1.64) | 1.98 (1.57)
  24 hours: number analyzed (Participants) | 2 | 4 | 1 | 2
  24 hours | 0.69 (1.42) | 1.92 (1.53) | 1.77 (1.71) | 2.00 (1.58)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 15 minutes; Test type: Superiority or Other; p = 0.034, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [0.02 to 0.57]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 15 minutes; Test type: Superiority or Other; p = 0.111, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.05 to 0.49]
Statistical Analysis 3: Comparison: Placebo vs Naproxen; 15 minutes; Test type: Superiority or Other; p = 0.125, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.06 to 0.48]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 30 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.81, 95% CI 2-sided [0.41 to 1.22]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 30 minutes; Test type: Superiority or Other; p = 0.003, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.61, 95% CI 2-sided [0.22 to 1.01]
Statistical Analysis 6: Comparison: Placebo vs Naproxen; 30 minutes; Test type: Superiority or Other; p = 0.004, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.59, 95% CI 2-sided [0.19 to 0.98]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 45 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.41, 95% CI 2-sided [0.91 to 1.91]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 45 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.24, 95% CI 2-sided [0.75 to 1.74]
Statistical Analysis 9: Comparison: Placebo vs Naproxen; 45 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.90, 95% CI 2-sided [0.41 to 1.39]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 60 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.63, 95% CI 2-sided [1.11 to 2.16]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 60 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.57, 95% CI 2-sided [1.05 to 2.09]
Statistical Analysis 12: Comparison: Placebo vs Naproxen; 60 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.26, 95% CI 2-sided [0.75 to 1.78]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 90 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.99, 95% CI 2-sided [1.46 to 2.52]
Statistical Analysis 14: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 90 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.09, 95% CI 2-sided [1.57 to 2.61]
Statistical Analysis 15: Comparison: Placebo vs Naproxen; 90 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.68, 95% CI 2-sided [1.16 to 2.20]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 2 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.12, 95% CI 2-sided [1.59 to 2.64]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 2 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.22, 95% CI 2-sided [1.70 to 2.74]
Statistical Analysis 18: Comparison: Placebo vs Naproxen; 2 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.69, 95% CI 2-sided [1.18 to 2.21]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 3 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.50, 95% CI 2-sided [1.98 to 3.01]
Statistical Analysis 20: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 3 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.48, 95% CI 2-sided [1.97 to 2.99]
Statistical Analysis 21: Comparison: Placebo vs Naproxen; 3 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.88, 95% CI 2-sided [1.37 to 2.38]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 4 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.54, 95% CI 2-sided [2.01 to 3.07]
Statistical Analysis 23: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 4 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.45, 95% CI 2-sided [1.92 to 2.97]
Statistical Analysis 24: Comparison: Placebo vs Naproxen; 4 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.81, 95% CI 2-sided [1.29 to 2.33]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 5 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.47, 95% CI 2-sided [1.92 to 3.03]
Statistical Analysis 26: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 5 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.41, 95% CI 2-sided [1.87 to 2.96]
Statistical Analysis 27: Comparison: Placebo vs Naproxen; 5 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.71, 95% CI 2-sided [1.16 to 2.25]
Statistical Analysis 28: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 6 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.26, 95% CI 2-sided [1.69 to 2.83]
Statistical Analysis 29: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 6 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.37, 95% CI 2-sided [1.80 to 2.93]
Statistical Analysis 30: Comparison: Placebo vs Naproxen; 6 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.67, 95% CI 2-sided [1.11 to 2.23]
Statistical Analysis 31: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 7 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.22, 95% CI 2-sided [1.66 to 2.79]
Statistical Analysis 32: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 7 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.30, 95% CI 2-sided [1.74 to 2.85]
Statistical Analysis 33: Comparison: Placebo vs Naproxen; 7 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.57, 95% CI 2-sided [1.02 to 2.13]
Statistical Analysis 34: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 8 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.19, 95% CI 2-sided [1.59 to 2.78]
Statistical Analysis 35: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 8 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.12, 95% CI 2-sided [1.53 to 2.70]
Statistical Analysis 36: Comparison: Placebo vs Naproxen; 8 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.63, 95% CI 2-sided [1.04 to 2.21]
Statistical Analysis 37: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 9 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.91, 95% CI 2-sided [1.30 to 2.52]
Statistical Analysis 38: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 9 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.12, 95% CI 2-sided [1.52 to 2.72]
Statistical Analysis 39: Comparison: Placebo vs Naproxen; 9 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.51, 95% CI 2-sided [0.91 to 2.11]
Statistical Analysis 40: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 10 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.94, 95% CI 2-sided [1.34 to 2.55]
Statistical Analysis 41: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 10 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.19, 95% CI 2-sided [1.59 to 2.79]
Statistical Analysis 42: Comparison: Placebo vs Naproxen; 10 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.56, 95% CI 2-sided [0.97 to 2.16]
Statistical Analysis 43: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 11 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.90, 95% CI 2-sided [1.28 to 2.52]
Statistical Analysis 44: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 11 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.13, 95% CI 2-sided [1.52 to 2.75]
Statistical Analysis 45: Comparison: Placebo vs Naproxen; 11 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.59, 95% CI 2-sided [0.98 to 2.20]
Statistical Analysis 46: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 12 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.90, 95% CI 2-sided [1.26 to 2.54]
Statistical Analysis 47: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 12 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.03, 95% CI 2-sided [1.39 to 2.66]
Statistical Analysis 48: Comparison: Placebo vs Naproxen; 12 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.44, 95% CI 2-sided [0.81 to 2.07]
Statistical Analysis 49: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 13 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.83, 95% CI 2-sided [1.17 to 2.49]
Statistical Analysis 50: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 13 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.78, 95% CI 2-sided [1.13 to 2.43]
Statistical Analysis 51: Comparison: Placebo vs Naproxen; 13 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.42, 95% CI 2-sided [0.78 to 2.07]
Statistical Analysis 52: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 14 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.64, 95% CI 2-sided [0.95 to 2.32]
Statistical Analysis 53: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 14 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.61, 95% CI 2-sided [0.94 to 2.29]
Statistical Analysis 54: Comparison: Placebo vs Naproxen; 14 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.38, 95% CI 2-sided [0.71 to 2.06]
Statistical Analysis 55: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 16 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.58, 95% CI 2-sided [0.88 to 2.27]
Statistical Analysis 56: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 16 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.42, 95% CI 2-sided [0.73 to 2.10]
Statistical Analysis 57: Comparison: Placebo vs Naproxen; 16 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.40, 95% CI 2-sided [0.72 to 2.08]
Statistical Analysis 58: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 24 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.25, 95% CI 2-sided [0.53 to 1.96]
Statistical Analysis 59: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 24 hours; Test type: Superiority or Other; p = 0.003, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.08, 95% CI 2-sided [0.38 to 1.79]
Statistical Analysis 60: Comparison: Placebo vs Naproxen; 24 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.32, 95% CI 2-sided [0.61 to 2.02]

16. Secondary Outcome: Pain Relief Combined With Pain Intensity Difference (PRID) Score
Description: PRID=PID+PR, where PID: 4-point categorical pain intensity difference scale, 0 (none) to 3 (severe), score derived by subtracting postdose score from baseline and could range from -1 to 3. Baseline pain intensity score of at least 2 was required for study enrollment. Higher positive PID values indicated improvement. PR: 5-point categorical pain relief scale (None [0], A Little [1], Some [2], A Lot [3], Complete [4]). PRID score could range from -1 to 7 where higher scores indicated better pain relief and decrease in pain intensity.
Time Frame: 15, 30, 45, 60, 90 minutes and 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 16, and 24 hours
Population: ITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen IR/ER (Roller Compaction) | Ibuprofen IR/ER (Wet Granulation) | Naproxen
Number analyzed (Participants) | 29 | 53 | 56 | 58
units on a scale
  15 minutes | -0.07 (0.59) | 0.45 (1.08) | 0.38 (0.84) | 0.33 (0.80)
  30 minutes | 0.07 (1.00) | 1.42 (1.60) | 1.16 (1.40) | 1.09 (1.37)
  45 minutes | 0.21 (1.08) | 2.49 (2.04) | 2.25 (1.90) | 1.74 (1.58)
  60 minutes | 0.31 (1.14) | 2.98 (2.18) | 2.98 (1.90) | 2.48 (1.86)
  90 minutes | 0.34 (1.20) | 3.64 (2.22) | 3.79 (1.92) | 3.14 (1.88)
  2 hours: number analyzed (Participants) | 13 | 51 | 54 | 53
  2 hours | 0.55 (1.45) | 4.17 (2.08) | 4.25 (1.97) | 3.29 (1.91)
  3 hours: number analyzed (Participants) | 8 | 51 | 53 | 52
  3 hours | 0.55 (1.92) | 4.75 (1.94) | 4.68 (1.87) | 3.67 (2.03)
  4 hours: number analyzed (Participants) | 7 | 51 | 51 | 51
  4 hours | 0.66 (2.13) | 4.98 (1.80) | 4.73 (1.97) | 3.67 (2.15)
  5 hours: number analyzed (Participants) | 7 | 51 | 51 | 50
  5 hours | 0.72 (2.14) | 4.87 (1.83) | 4.75 (2.08) | 3.59 (2.32)
  6 hours: number analyzed (Participants) | 7 | 51 | 51 | 47
  6 hours | 0.79 (2.21) | 4.60 (1.96) | 4.75 (2.06) | 3.62 (2.35)
  7 hours: number analyzed (Participants) | 7 | 51 | 51 | 47
  7 hours | 0.79 (2.21) | 4.45 (1.90) | 4.66 (2.08) | 3.41 (2.32)
  8 hours: number analyzed (Participants) | 7 | 49 | 50 | 46
  8 hours | 0.72 (2.10) | 4.30 (1.95) | 4.25 (2.30) | 3.41 (2.35)
  9 hours: number analyzed (Participants) | 7 | 49 | 50 | 45
  9 hours | 0.66 (1.95) | 3.89 (2.14) | 4.18 (2.29) | 3.16 (2.36)
  10 hours: number analyzed (Participants) | 7 | 47 | 50 | 44
  10 hours | 0.55 (1.82) | 3.77 (2.19) | 4.21 (2.38) | 3.16 (2.38)
  11 hours: number analyzed (Participants) | 7 | 46 | 49 | 44
  11 hours | 0.55 (1.94) | 3.70 (2.22) | 4.14 (2.39) | 3.21 (2.50)
  12 hours: number analyzed (Participants) | 7 | 46 | 47 | 41
  12 hours | 0.52 (1.92) | 3.70 (2.24) | 3.95 (2.45) | 2.93 (2.53)
  13 hours: number analyzed (Participants) | 6 | 43 | 44 | 41
  13 hours | 0.62 (2.03) | 3.68 (2.39) | 3.63 (2.59) | 2.98 (2.46)
  14 hours: number analyzed (Participants) | 6 | 41 | 43 | 40
  14 hours | 0.69 (2.17) | 3.43 (2.51) | 3.45 (2.68) | 2.97 (2.54)
  16 hours: number analyzed (Participants) | 6 | 39 | 39 | 38
  16 hours | 0.55 (2.01) | 3.23 (2.43) | 3.02 (2.67) | 2.93 (2.57)
  24 hours: number analyzed (Participants) | 2 | 4 | 1 | 2
  24 hours | 0.76 (2.34) | 2.81 (2.45) | 2.68 (2.78) | 2.97 (2.58)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 15 minutes; Test type: Superiority or Other; p = 0.011, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [0.12 to 0.91]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 15 minutes; Test type: Superiority or Other; p = 0.028, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [0.05 to 0.83]
Statistical Analysis 3: Comparison: Placebo vs Naproxen; 15 minutes; Test type: Superiority or Other; p = 0.048, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [0.00 to 0.78]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 30 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.32, 95% CI 2-sided [0.69 to 1.96]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 30 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.08, 95% CI 2-sided [0.45 to 1.71]
Statistical Analysis 6: Comparison: Placebo vs Naproxen; 30 minutes; Test type: Superiority or Other; p = 0.002, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.01, 95% CI 2-sided [0.38 to 1.63]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 45 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.26, 95% CI 2-sided [1.46 to 3.06]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 45 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.03, 95% CI 2-sided [1.24 to 2.82]
Statistical Analysis 9: Comparison: Placebo vs Naproxen; 45 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.52, 95% CI 2-sided [0.74 to 2.31]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 60 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.64, 95% CI 2-sided [1.78 to 3.50]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 60 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.66, 95% CI 2-sided [1.81 to 3.51]
Statistical Analysis 12: Comparison: Placebo vs Naproxen; 60 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.16, 95% CI 2-sided [1.32 to 3.00]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 90 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.26, 95% CI 2-sided [2.39 to 4.12]
Statistical Analysis 14: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 90 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.42, 95% CI 2-sided [2.57 to 4.28]
Statistical Analysis 15: Comparison: Placebo vs Naproxen; 90 minutes; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.77, 95% CI 2-sided [1.92 to 3.63]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 2 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.57, 95% CI 2-sided [2.70 to 4.44]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 2 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.68, 95% CI 2-sided [2.82 to 4.53]
Statistical Analysis 18: Comparison: Placebo vs Naproxen; 2 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.72, 95% CI 2-sided [1.87 to 3.57]
Statistical Analysis 19: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 3 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 4.13, 95% CI 2-sided [3.27 to 4.99]
Statistical Analysis 20: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 3 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 4.09, 95% CI 2-sided [3.24 to 4.95]
Statistical Analysis 21: Comparison: Placebo vs Naproxen; 3 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.09, 95% CI 2-sided [2.24 to 3.93]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 4 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 4.25, 95% CI 2-sided [3.36 to 5.13]
Statistical Analysis 23: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 4 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 4.04, 95% CI 2-sided [3.17 to 4.92]
Statistical Analysis 24: Comparison: Placebo vs Naproxen; 4 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.98, 95% CI 2-sided [2.11 to 3.85]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 5 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 4.07, 95% CI 2-sided [3.14 to 5.01]
Statistical Analysis 26: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 5 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 4.00, 95% CI 2-sided [3.07 to 4.92]
Statistical Analysis 27: Comparison: Placebo vs Naproxen; 5 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.83, 95% CI 2-sided [1.91 to 3.75]
Statistical Analysis 28: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 6 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.75, 95% CI 2-sided [2.78 to 4.71]
Statistical Analysis 29: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 6 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.93, 95% CI 2-sided [2.98 to 4.89]
Statistical Analysis 30: Comparison: Placebo vs Naproxen; 6 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.80, 95% CI 2-sided [1.85 to 3.75]
Statistical Analysis 31: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 7 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.61, 95% CI 2-sided [2.65 to 4.56]
Statistical Analysis 32: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 7 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.84, 95% CI 2-sided [2.89 to 4.79]
Statistical Analysis 33: Comparison: Placebo vs Naproxen; 7 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.60, 95% CI 2-sided [1.65 to 3.54]
Statistical Analysis 34: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 8 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.54, 95% CI 2-sided [2.54 to 4.53]
Statistical Analysis 35: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 8 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.51, 95% CI 2-sided [2.52 to 4.49]
Statistical Analysis 36: Comparison: Placebo vs Naproxen; 8 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.67, 95% CI 2-sided [1.69 to 3.65]
Statistical Analysis 37: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 9 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.20, 95% CI 2-sided [2.19 to 4.21]
Statistical Analysis 38: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 9 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.51, 95% CI 2-sided [2.51 to 4.51]
Statistical Analysis 39: Comparison: Placebo vs Naproxen; 9 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.49, 95% CI 2-sided [1.49 to 3.48]
Statistical Analysis 40: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 10 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.19, 95% CI 2-sided [2.17 to 4.21]
Statistical Analysis 41: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 10 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.65, 95% CI 2-sided [2.64 to 4.66]
Statistical Analysis 42: Comparison: Placebo vs Naproxen; 10 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.59, 95% CI 2-sided [1.58 to 3.60]
Statistical Analysis 43: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 11 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.10, 95% CI 2-sided [2.06 to 4.15]
Statistical Analysis 44: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 11 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.57, 95% CI 2-sided [2.53 to 4.61]
Statistical Analysis 45: Comparison: Placebo vs Naproxen; 11 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.64, 95% CI 2-sided [1.61 to 3.67]
Statistical Analysis 46: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 12 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.15, 95% CI 2-sided [2.09 to 4.21]
Statistical Analysis 47: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 12 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.41, 95% CI 2-sided [2.36 to 4.46]
Statistical Analysis 48: Comparison: Placebo vs Naproxen; 12 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.40, 95% CI 2-sided [1.36 to 3.44]
Statistical Analysis 49: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 13 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 3.03, 95% CI 2-sided [1.94 to 4.12]
Statistical Analysis 50: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 13 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.99, 95% CI 2-sided [1.91 to 4.07]
Statistical Analysis 51: Comparison: Placebo vs Naproxen; 13 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.35, 95% CI 2-sided [1.28 to 3.42]
Statistical Analysis 52: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 14 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.70, 95% CI 2-sided [1.57 to 3.83]
Statistical Analysis 53: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 14 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.74, 95% CI 2-sided [1.62 to 3.85]
Statistical Analysis 54: Comparison: Placebo vs Naproxen; 14 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.26, 95% CI 2-sided [1.14 to 3.37]
Statistical Analysis 55: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 16 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.64, 95% CI 2-sided [1.51 to 3.76]
Statistical Analysis 56: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 16 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.45, 95% CI 2-sided [1.33 to 3.56]
Statistical Analysis 57: Comparison: Placebo vs Naproxen; 16 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.36, 95% CI 2-sided [1.25 to 3.47]
Statistical Analysis 58: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); 24 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.02, 95% CI 2-sided [0.86 to 3.19]
Statistical Analysis 59: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); 24 hours; Test type: Superiority or Other; p = 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 1.90, 95% CI 2-sided [0.75 to 3.05]
Statistical Analysis 60: Comparison: Placebo vs Naproxen; 24 hours; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.19, 95% CI 2-sided [1.05 to 3.34]

17. Secondary Outcome: Peak Pain Relief Score
Description: Maximum PR score over the scheduled pain relief assessments. PR score based on 5-point categorical pain relief scale. Participants asked, "How much relief do you have from your starting pain?" Range of scale: None (0), A Little (1), Some (2), A Lot (3) or Complete (4). Higher scores indicated improvement (better pain relief).
Time Frame: Baseline to 12 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen IR/ER (Roller Compaction) | Ibuprofen IR/ER (Wet Granulation) | Naproxen
Number analyzed (Participants) | 29 | 53 | 56 | 58
units on a scale | 1.00 (1.41) | 3.42 (0.82) | 3.39 (0.85) | 3.05 (1.16)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen IR/ER (Roller Compaction); Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.42, 95% CI 2-sided [1.94 to 2.89]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen IR/ER (Wet Granulation); Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.39, 95% CI 2-sided [1.92 to 2.86]
Statistical Analysis 3: Comparison: Placebo vs Naproxen; Test type: Superiority or Other; p < 0.001, ANOVA — p-value adjusted for baseline PSR and gender; Mean Difference (Final Values) = 2.05, 95% CI 2-sided [1.58 to 2.52]

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another subject, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | Ibuprofen IR/ER (Roller Compaction) | Ibuprofen IR/ER (Wet Granulation) | Naproxen
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/53 | 0/56 | 0/58
Other Adverse Events (participants affected / at risk) | 8/29 | 3/53 | 8/56 | 6/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | Ibuprofen IR/ER (Roller Compaction) (N=53) | Ibuprofen IR/ER (Wet Granulation) (N=56) | Naproxen (N=58)
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 1 | 5 | 2
Vomiting (Gastrointestinal disorders) | 5 | 0 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 2
Headache (Nervous system disorders) | 1 | 2 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Epistaxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.